CLINICAL TRIAL: NCT01528397
Title: Reconstruction of Proper Digital Nerve Defects in the Thumb Using a Pedicled Nerve Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Hospital of Tangshan (Other)
Collaborators: Chinese PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TSChen3885
Record Dates: First submitted 2012-01-31; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-01

CONDITIONS: Nerve Injury
Keywords: defect; dorsal branch of the proper digital nerve; proper digital nerve; second dorsal metacarpal artery; pedicled nerve graft.

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: pedicled nerve graft — A pedicled nerve graft harvested from the dorsal branch of the PDN can be used for reconstruction of such defects. The graft is based on the second dorsal metacarpal artery.
  Other Names: Vascularized nerve graft

SUMMARY:
A proper digital nerve (PDN) defect in the thumb can produce partial or complete sensory loss which can result in functional disability. This article reports the treatment of the thumb PDN defect using a pedicled nerve graft harvested from the dorsal branch of the PDN. Fourteen patients with the thumb PDN defect underwent a new surgical procedure in which the pedicled nerve graft was used to bridge nerve defect. For comparison, the investigators also collected a consecutive series of 21 patients with thumb PDN defects treated using a nonvascularized sural nerve graft. This study was designed to evaluate the efficacy of pedicled nerve grafting for PDN defects in the thumb.

DETAILED DESCRIPTION:
At final follow-up, the investigators measured the sensibility of the thumb pulps and the donor sites using the Semmes-Weinstein monofilament test and static 2-point discrimination (2PD) test. The test points were at the centers of the radial and ulnar portions of the thumb pulp and the donor sites separately. Each area was tested 3 times with a Dellon-Mackinnon discriminator. Two out of 3 correct answers were considered proof of perception before proceeding to another lower value.

ELIGIBILITY:
Inclusion Criteria:

1. thumb PDN defects between the middle of the distal phalanx and the metacarpophalangeal joint;
2. PDN defects of single or both sides;
3. PDN defects 1-4 cm in length.

Exclusion Criteria:

1. injury to the course of the pedicle or the donor sites;
2. PDN defects less than 1 cm or longer than 4 cm;
3. no Doppler sound at the location of the second dorsal metacarpal artery (SDMA).

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
static 2-point discrimination (2PD) test | 22 months
  The test points were at the centers of the radial and ulnar portions of the thumb pulp and the donor sites separately. Each area was tested 3 times with a Dellon-Mackinnon discriminator. Two out of 3 correct answers were considered proof of perception before proceeding to another lower value.

REFERENCES:
- [Derived] Chen C, Tang P, Zhang X. Reconstruction of proper digital nerve defects in the thumb using a pedicle nerve graft. Plast Reconstr Surg. 2012 Nov;130(5):1089-1097. doi: 10.1097/PRS.0b013e318267d56b. PMID 23096609